CLINICAL TRIAL: NCT03449680
Title: The Analgesic Efficacy of the Ultrasound-Guided Femoral Articular Branch Block for Ambulatory Hip Arthroscopy: A Randomized-Controlled Trial
Brief Title: The Analgesic Efficacy of the Ultrasound-Guided Femoral Articular Branch Block for Ambulatory Hip Arthroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Women's College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016-0119-B
Record Dates: First submitted 2017-09-01; First posted 2018-02-28 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Anesthesia, Regional
Keywords: hip arthroscopy; femoral articular branch block

STUDY DESIGN:
Intervention Model Description: Patients will be randomized between one of two treatment groups. The intervention of femoral articular branch block or the control group (non-invasive placebo).
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The anesthesiologist performing the nerve block will be aware of group allocation; but a separate anesthesiologist providing intra-operative care will remain blinded. The patient and the research staff collecting outcome data will remain blinded until all data are collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Femoral Articular Branch Block (Experimental): Patients will receive an ultrasound-guided femoral articular branch block with an injection of 20ml of ropivicaine 0.5%
  Interventions: Procedure: Femoral Articular Branch Block
- Placebo Block (Placebo Comparator): Patients will receive an ultrasound simulation of the location of a femoral articular branch block , this is to maintain blinding. A subcutaneous injection of 1ml of normal sterile saline will be administered
  Interventions: Procedure: Placebo Block

INTERVENTIONS:
Procedure: Femoral Articular Branch Block — Slow injection (3mL aliquots) of local anesthetic solution (20ml of Ropivacaine 0.5%) into the fascia above the iliopsoas muscle (located in the groove between the two bony landmarks - (1)anterior inferior iliac crest and (2)iliopubic eminence).This is done by ultrasound guidance.
  Arms: Femoral Articular Branch Block
Procedure: Placebo Block — Subcutaneous injection of 1ml normal sterile saline
  Arms: Placebo Block

SUMMARY:
Hip arthroscopy surgery can be associated with significant pain. A regional anesthesia technique, the femoral articular branch block (FAB), has recently been proposed to collectively block terminal femoral and accessory obturator nerve branches to the hip joint with a single injection, theoretically blocking most of the innervation relevant to hip arthroscopy while sparing the main femoral nerve branches to the quadriceps muscles. The investigators aim to demonstrate the analgesic benefits of FAB. The investigators hypothesize that FAB will reduce opioid consumption and improve postoperative quality of recovery in patients having hip arthroscopy. This is a randomized, controlled, double-blind study and half the patients will be randomized to receive the femoral articular branch block and the other half of patients will be randomized to receive a placebo block. A comparison of pain will be made between both groups.

DETAILED DESCRIPTION:
Hip arthroscopy is a surgical technique that is gaining popularity for its diagnostic and therapeutic role in the management of adult hip pain. This procedure is frequently associated with severe post-operative pain despite the practice of injecting the hip joint with local anesthetics at the end of the procedure and the use of intraoperative opioids. The ideal analgesic technique that provides adequate pain relief following this procedure has not been established yet.

There is evidence to suggest that a femoral nerve block (FNB) may provide clinically meaningful analgesia. The investigators have examined the benefits of FNB both retrospectively and prospectively in hip arthroscopy patients at Women's College Hospital (WCH). Both of our studies suggested modest benefits of the FNB in terms of controlling post-operative pain and reducing opioid consumption. However the majority of patients continued to experience moderate to severe post-operative pain and required significant amounts of opioid analgesics in the Peri-Anesthesia Unit (PAU), despite receiving the FNB.

Another regional anesthesia technique, the femoral articular branch block (FAB) has recently been proposed to collectively block the terminal femoral and accessory obturator nerve branches to the hip joint with a single injection, theoretically blocking most of the innervation relevant to hip arthroscopy while sparing the main femoral nerve branches to the quadriceps muscle. The investigators aim to demonstrate the analgesic benefits of FAB.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical classification system, ASA I-III patients
* 18 - 60 years of age
* Body Mass Index (BMI) <35 kg/m2

Exclusion Criteria:

* Pre-existing neurological deficits or peripheral neuropathy in the distribution of femoral, obturator, or lateral cutaneous nerves
* Local infection
* Contra-indication to regional anesthesia e.g. bleeding diathesis, coagulopathy
* Chronic pain disorders
* History of using over 30mg of oxycodone or equivalent per day
* Contraindication to a component of multi-modal analgesia
* Allergy to local anesthesia
* History of significant psychiatric conditions that may affect patient assessment
* Pregnancy
* Inability to provide informed consent
* Patient refusal of femoral articular branch block
* Revision arthroscopy surgeries

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2018-03-04 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Analgesic Consumption | 24 hours postoperatively
  Postoperative cumulative oral morphine equivalent consumption during the first 24 hours will be the first primary outcome
Quality of Life scores | 24 hours postoperatively
  Quality of Recovery (QR15) scores at 24 hours will be the second primary outcome.
  QR15 is a measurement of quality of recovery after surgery and anesthesia that has been psychometrically tested and validated. Reporting of outcome measures on a scale of 0 to 10 (0=None of the time and 10=All of the time). There are a total of 40 items/questions.

SECONDARY OUTCOMES:
Pain Assessment (VAS) | Up to 48 hours post-operatively and at 7-day mark
  Visual Analogue Scale(VAS) - Pain:Overall pain assessed at rest and on movement A continuous scale comprised of a 100mm (10cm) horizontal line, anchored by 2 verbal descriptions No Pain to Worst Pain
Analgesic Consumption | Up to 48 hours following surgery
  Consumption intra-operatively, total in-hospital postoperative consumption, and time to first analgesic request in the first 24 hours, cumulative oral morphine equivalent
Presence of Block-related complications | Up until one month following nerve block
  vascular puncture, hematoma formation, intravascular injection, epidural anesthesia-bilateral sensory block Presence/ absence of residual paresthesia or numbness over femoral, obturator, and lateral cutaneous nerves distribution
Incidence of opioid-related side effects | Up until one month following nerve block
  nausea, vomiting, pruritus, sedation
Patient Satisfaction with Analgesic Technique | One month after surgery
  A Patient Diary will be completed to assess overall satisfaction with analgesic technique
Demographic Data | Day 1 - first 24 hours
  Patient demographics - There is no scale, just questions asked of the participant.
Turn over time | after surgery up to discharge, assessed up to 24 hours
  PAU leaving time

CONTACTS AND LOCATIONS:
Overall Officials: Richard Brull, MD, Principal Investigator — Women's College Hospital, University of Toronto; Daniel Whelan, MD, Principal Investigator — Women's College Hospital, University of Toronto
Locations (1):
- Women's College Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Short AJ, Barnett JJG, Gofeld M, Baig E, Lam K, Agur AMR, Peng PWH. Anatomic Study of Innervation of the Anterior Hip Capsule: Implication for Image-Guided Intervention. Reg Anesth Pain Med. 2018 Feb;43(2):186-192. doi: 10.1097/AAP.0000000000000701. PMID 29140962
- [Result] Suzuki S, Awaya G, Okada Y, Maekawa M, Ikeda T, Tada H. Arthroscopic diagnosis of ruptured acetabular labrum. Acta Orthop Scand. 1986 Dec;57(6):513-5. doi: 10.3109/17453678609014781. PMID 3577718
- [Result] Larson CM, Swaringen J, Morrison G. A review of hip arthroscopy and its role in the management of adult hip pain. Iowa Orthop J. 2005;25:172-9. PMID 16089093
- [Result] Baber YF, Robinson AH, Villar RN. Is diagnostic arthroscopy of the hip worthwhile? A prospective review of 328 adults investigated for hip pain. J Bone Joint Surg Br. 1999 Jul;81(4):600-3. doi: 10.1302/0301-620x.81b4.8803. PMID 10463728
- [Result] Lee EM, Murphy KP, Ben-David B. Postoperative analgesia for hip arthroscopy: combined L1 and L2 paravertebral blocks. J Clin Anesth. 2008 Sep;20(6):462-5. doi: 10.1016/j.jclinane.2008.04.012. PMID 18929290
- [Result] Baker JF, Byrne DP, Hunter K, Mulhall KJ. Post-operative opiate requirements after hip arthroscopy. Knee Surg Sports Traumatol Arthrosc. 2011 Aug;19(8):1399-402. doi: 10.1007/s00167-010-1248-4. Epub 2010 Sep 9. PMID 20827460
- [Result] Ward JP, Albert DB, Altman R, Goldstein RY, Cuff G, Youm T. Are femoral nerve blocks effective for early postoperative pain management after hip arthroscopy? Arthroscopy. 2012 Aug;28(8):1064-9. doi: 10.1016/j.arthro.2012.01.003. Epub 2012 Apr 11. PMID 22498045
- [Result] Dold AP, Murnaghan L, Xing J, Abdallah FW, Brull R, Whelan DB. Preoperative femoral nerve block in hip arthroscopic surgery: a retrospective review of 108 consecutive cases. Am J Sports Med. 2014 Jan;42(1):144-9. doi: 10.1177/0363546513510392. Epub 2013 Nov 27. PMID 24284048
- [Result] Xing JG, Abdallah FW, Brull R, Oldfield S, Dold A, Murnaghan ML, Whelan DB. Preoperative Femoral Nerve Block for Hip Arthroscopy: A Randomized, Triple-Masked Controlled Trial. Am J Sports Med. 2015 Nov;43(11):2680-7. doi: 10.1177/0363546515602468. Epub 2015 Sep 24. PMID 26403206
- [Result] GARDNER E. The innervation of the hip joint. Anat Rec. 1948 Jul;101(3):353-71. doi: 10.1002/ar.1091010309. No abstract available. PMID 18873153
- [Result] Dee R. Structure and function of hip joint innervation. Ann R Coll Surg Engl. 1969 Dec;45(6):357-74. No abstract available. PMID 5359432
- [Result] Birnbaum K, Prescher A, Hessler S, Heller KD. The sensory innervation of the hip joint--an anatomical study. Surg Radiol Anat. 1997;19(6):371-5. doi: 10.1007/BF01628504. PMID 9479711